CLINICAL TRIAL: NCT00875706
Title: Training and Coaching to Promote High Performance in VA Nursing Home Care
Brief Title: Training and Coaching to Promote High Performance in Veteran Affairs (VA) Nursing Home Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None | Purpose: Health Services Research
Other Study IDs: EDU 08-427
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Dementia
Keywords: Nursing Homes; Implementation of innovative programs; Nursing staff; Nurses' aides; Educational models
MeSH Terms: conditions — Dementia | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training Feasibility (Other): 4 sites will receive the training intervention to determine the feasibility of the train-the trainer approach.
  The educational intervention is included in this arm.
  Interventions: Behavioral: Educational Intervention
- Data Collection - Survey (Other): Survey data collection tools will be piloted to assess feasibility of survey administration and development of the survey for future studies. This tools were piloted in sites where the educational intervention was administered.
  Interventions: Behavioral: Educational Intervention
- Data Collection - Interview (Other): Interview data collection tools will be piloted to assess feasibility of interview administration and development of the interview protocol for future studies. This tools were piloted in sites where the educational intervention was administered.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — The intervention consists of two (2) different types of training, both to be delivered through a train-the-trainer approach. The first of these is coaching-supervision training for nurse managers and other supervisory personnel in the CLC units. The second component is a one-day training for DCWs on communication and managing problem behaviors associated with dementia. These two trainings build on validated training models that have been developed by PHINational, but will be adapted and customized to include VA-developed clinical content on the management of problem behaviors associated with dementia.

SUMMARY:
This study aimed to explore the feasibility of an educational intervention to strengthen workplace learning systems in four VA Community Living Centers (CLCs).

DETAILED DESCRIPTION:
Background:

The study explored the feasibility of an educational intervention to strengthen workplace-learning systems in four VA Community Living Centers (CLCs).

Objectives:

Specific aims were to 1) conduct a feasibility study to assess whether the educational intervention is practical to implement as designed and 2) conduct a pilot study to validate the methodology proposed for assessing outcomes of this educational intervention.

Methods:

A multi-level intervention targeting the translation of workplace learning into practice was implemented. The Direct Care Worker (DCW) intervention targeted both clinical knowledge and effective communication. The Coaching Supervision training addressed management and supervision practices for nurses, combined with effective communication. Four CLCs received both interventions, administered by the Paraprofessional Health Institute (PHI), using a train-the-trainer approach over the course of four 3-day sessions. Quantitative and qualitative data were collected to assess factors influencing effectiveness of implementation and to understand the impact of the trainings on participants.

Status:

The study has been completed with educational interventions implemented and qualitative and quantitative data collected.

ELIGIBILITY:
Inclusion Criteria:

* VA Employees: psychologists, nurse-managers and front-line nursing care staff assigned to CLCs will be included

Exclusion Criteria:

* Those not working in the CLC,
* Those working in the CLC but not involved in the training intervention that is the focus of the study (e.g. Environment Management Service personnel, dietary personnel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol VanDeusen-Lukas, EdD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Training Feasibility: 4 sites (8 individuals) received the training intervention to determine the feasibility of the train-the trainer approach.
  The educational intervention is included in this arm.
  Educational Intervention: The intervention consists of two (2) different types of training, both to be delivered through a train-the-trainer approach. The first of these is coaching-supervision training for nurse managers and other supervisory personnel in the CLC units. The second component is a one-day training for DCWs on communication and managing problem behaviors associated with dementia. These two trainings build on validated training models that have been developed by PHINational, but will be adapted and customized to include VA-developed clinical content on the management of problem behaviors associated with dementia.
- Data Collection - Survey: Survey data collection tools were piloted to assess feasibility of survey administration and development for use in a long-term care setting. These tools were piloted in sites where the educational intervention was administered.
  The survey was a modified version of the Care Coordination Survey which was originally validated in a hospital setting (citation below). The survey pertains to work context factors that shape practice, including staffing and resources, communication and IT, participation in decision-making, relationships with supervisors, professional empowerment, and relational coordination. Modifications were made for use of the survey in a VA Community Living Centers.
  Weinberg, D., J. Perloff, D. Cooney-Miner, and E. Glaser, Supporting work and workers: Validation of a hospital work organization survey for professional and paraprofessional workers. 2008.
- Data Collection - Interview: Interview data collection tools were piloted to assess feasibility of interview administration and development of the interview protocol for future studies. These tools were piloted in sites where the educational intervention was administered.
Period: Overall Study
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview
Started | 8 | 24 | 13
Completed | 7 | 24 | 13
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Training Feasibility: 4 sites (8 individuals) received the training intervention to determine the feasibility of the train-the trainer approach.
  The educational intervention is included in this arm.
- Data Collection - Survey: Survey data collection tools were piloted to assess feasibility of survey administration and development of the survey for future studies. These tools were piloted in sites where the educational intervention was administered.
- Total: Total of all reporting groups
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview | Total
Number analyzed (Participants) | 8 | 24 | 13 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Age was not collected as it was not pertinent to the study. | NA — Age was not collected as it was not pertinent to the study. | NA — Age was not collected as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — Age was not collected as it was not pertinent to the study. | NA — Age was not collected as it was not pertinent to the study. | NA — Age was not collected as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Age was not collected as it was not pertinent to the study. | NA — Age was not collected as it was not pertinent to the study. | NA — Age was not collected as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Number; unit: participants]
  Male | NA — Gender was not collected for this portion of the study as it was not pertinent to the study. | 4 | NA — Gender was not collected for this portion of the study as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Female | NA — Gender was not collected for this portion of the study as it was not pertinent to the study. | 19 | NA — Gender was not collected for this portion of the study as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown | NA — Gender was not collected for this portion of the study as it was not pertinent to the study. | 1 | NA — Gender was not collected for this portion of the study as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaskan Native | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | 0 | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | 0 | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | 5 | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian/Other Pacific Islander | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | 0 | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | 17 | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | 2 | NA — Race/Ethnicity was not collected for this Arm as it was not pertinent to the study. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Completion of Training Intervention
Description: This outcome measures the number of participants that fully completed the training intervention.
Time Frame: This outcome was assessed at the end of the 1 year pilot study.
Population: The analysis population includes only participants who started the Train-the-Trainer intervention and therefore only participants in the Training Feasibility Arm/Group were analyzed for this outcome.
Measure: Number; unit: participants
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview
Number analyzed (Participants) | 8 | 0 | 0
participants | 7 |  |

2. Primary Outcome: Facility Implementation of Trainings
Description: This measure assesses the number of participating facilities (4) that implemented trainings in their own facilities upon completion of our educational training intervention.
Time Frame: This outcome was assessed at the end of the 1 year pilot study.
Population: This unit of measure for this outcome measure is at the facility level. There were 4 facilities (8 trainees) in total that began the training intervention.
Measure: Number; unit: Facility
Units Other Than Participants: Facility
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview
Number analyzed (Participants) | 8 | 0 | 0
Number analyzed (Facility) | 4 | 0 | 0
Facility
  Coaching and Supervision Training | 3 |  |
  Direct Care Worker Training | 2 |  |

3. Primary Outcome: Number of Participants in Pilot Surveys
Description: This outcome measures the number of participants that completed the survey during the pilot in order to assess the feasibility of conducting a larger study.
Time Frame: This outcome was assessed at the end of the 1 year pilot study.
Population: Only participants in the Data Collection - Survey group were analyzed for this outcome. The population included trainees and direct care workers.
Measure: Number; unit: participants
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview
Number analyzed (Participants) | 0 | 24 | 0
participants |  | 24 |

4. Primary Outcome: Number of Participants in Pilot Interviews
Description: This outcome measures the number of participants that participated in interviews that were conducted during the pilot in order to assess the feasibility of conducting a larger study.
Time Frame: This outcome was assessed at the end of the 1 year pilot study.
Population: Only participants in the Data Collection - Interview group were analyzed for this outcome. The population included trainees and direct care workers.
Measure: Number; unit: participants
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview
Number analyzed (Participants) | 0 | 0 | 13
participants |  |  | 13

ADVERSE EVENTS:
Description: No serious or other adverse events were collected.
Arm/Group | Training Feasibility | Data Collection - Survey | Data Collection - Interview
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes